CLINICAL TRIAL: NCT01480258
Title: A Phase III Randomized, Double-Blind, Active-Comparator Controlled Clinical Trial to Study the Safety, Tolerability, and Immunogenicity of V419 in Healthy Infants When Given at 2, 4, and 11 to 12 Months
Brief Title: Safety, Tolerability, and Immunogenicity of V419 in Healthy Infants When Given at 2, 4, and 11 to 12 Months (V419-008)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MCM Vaccines B.V. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V419-008; 2010-021491-28 (EudraCT Number); V419-008 (Other: Merck)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Bacterial Infections; Virus Diseases
Keywords: combination vaccine; diphtheria; pertussis; tetanus; hepatitis B; Hep B; Haemophilus influenzae b; Hib; polio; poliovirus
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Diphtheria; Whooping Cough; Tetanus; Hepatitis B; Haemophilus Infections; Poliomyelitis | interventions — Vaxelis; Rotavirus Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PR5I (Experimental): Infant series: PR5I 0.5 mL injection + Prevenar 13™ 0.5 mL injection administered at 2 and 4 months of age, and rotavirus vaccine (either Rotarix™ 1.5 mL oral dose at 2 and 4 months of age [subset 1] or RotaTeq™ 2 mL oral dose at 2, 4 and 5 months of age [subset 2]).
  Toddler dose: PR5I 0.5 mL injection + Prevenar 13™ 0.5 mL injection administered at 11 to 12 months of age.
  Interventions: Biological: PR5I; Biological: Rotavirus vaccine; Biological: Prevenar 13™
- INFANRIX™ hexa (Active Comparator): Infant series: INFANRIX™ hexa 0.5 mL injection + Prevenar 13™ 0.5 mL injection administered at 2 and 4 months of age, and rotavirus vaccine (either Rotarix™ 1.5 mL oral dose at 2 and 4 months of age [subset 1] or RotaTeq™ 2 mL oral dose at 2, 4 and 5 months of age [subset 2]).
  Toddler dose: INFANRIX™ hexa 0.5 mL injection + Prevenar 13™ 0.5 mL injection administered at 11 to 12 months of age.
  Interventions: Biological: Rotavirus vaccine; Biological: Prevenar 13™; Biological: INFANRIX™ hexa

INTERVENTIONS:
Biological: PR5I — DTaP-HB-IPV-Hib (Diphtheria, tetanus, pertussis [acellular, component], hepatitis B [recombinant DNA], polio virus [inactivated], and Haemophilus influenza type b conjugate vaccine [adsorbed]) Vaccine 0.5 mL intramuscular injection at 2, 4, and 11 to 12 months of age. Injection is to be administered in the upper anterolateral thigh, separate limb from the concomitant vaccine. PR5I is a liquid suspension hexavalent vaccine.
  Other Names: V419; Vaxelis®
  Arms: PR5I
Biological: Rotavirus vaccine — Rotarix™ 1.5 mL oral dose at 2 and 4 months of age (subset 1, Italy and Sweden) or RotaTeq™ 2 mL oral dose at 2, 4 and 5 months of age (subset 2, Finland)
Biological: Prevenar 13™ — Prevenar 13™ 0.5 mL intramuscular injection at 2, 4, and 11 to 12 months of age. Injection is to be administered in the upper anterolateral thigh, separate limb from the concomitant vaccine.
Biological: INFANRIX™ hexa — Combined Diphtheria-Tetanus-acellular Pertussis [DTaP], Hepatitis B [HepB], Poliovirus [IPV] and Haemophilus influenzae type b [Hib] Vaccine 0.5 mL intramuscular injection at 2, 4 and 11 to 12 months of age. Injection is to be administered in the upper anterolateral thigh, separate limb from the concomitant vaccine. INFANRIX™ hexa is provided as 2 components (lyophilized Hib and liquid DTaP, IPV, and HepB). Prior to administration, the vaccine must be reconstituted by adding the liquid DTaP-HepB-IPV component to the vial containing the Hib pellet.
  Arms: INFANRIX™ hexa

SUMMARY:
This study will determine whether participants who receive V419 (PR5I) at 2, 4, and 11 to 12 months of age have an acceptable response to the vaccine. This study will also determine whether the immune response to V419 is similar to that of participants who received a licensed vaccine control. The primary hypothesis is that participants who receive PR5I at 2, 4, and 11 to 12 months have an acceptable response rate to all PR5I-contained antigens at one month after the Toddler dose of PR5I.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant able to attend all study visits
* Parent(s)/legal representative are able to read, understand, and complete study questionnaires

Exclusion Criteria:

* History of congenital or acquired immunodeficiency
* Received or is expected to receive immunosuppressive agents or systemic immunomodulatory steroids
* History of leukemia, lymphoma, malignant melanoma, or myeloproliferative disorder
* Hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances as the study vaccines or concomitant study vaccines
* Has any chronic illness that could interfere with study conduct or completion
* Received any immune globulin, blood, or blood-derived products since birth
* Received a dose of hepatitis B vaccine prior to study entry
* Vaccinated with any acellular pertussis or whole cell pertussis based combination vaccines, Haemophilus influenzae type b conjugate, poliovirus, pneumococcal conjugate or pneumococcal polysaccharide, rotavirus vaccine, or combination thereof
* Fever within 24 hours prior to enrollment
* Received any non-study vaccine within 30 days prior to enrollment, except for inactivated influenza vaccine, which is permitted 14 days or more prior to enrolment
* Has a coagulation disorder
* Has developmental delay or neurological disorder
* Participant or his/her mother has a medical history of hepatitis B surface antigens (HBsAg) seropositivity
* History of Haemophilus influenzae type b, hepatitis B, diphtheria, tetanus, pertussis, poliomyelitis, rotavirus gastroenteritis, or invasive pneumococcal infection

Ages: 46 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1315 (Actual)
Dates: Start 2011-11-23 (Actual); Primary Completion 2013-10-09 (Actual); Study Completion 2013-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Silfverdal SA, Icardi G, Vesikari T, Flores SA, Pagnoni MF, Xu J, Liu GF, Stek JE, Boisnard F, Thomas S, Ziani E, Lee AW. A Phase III randomized, double-blind, clinical trial of an investigational hexavalent vaccine given at 2, 4, and 11-12 months. Vaccine. 2016 Jul 19;34(33):3810-6. doi: 10.1016/j.vaccine.2016.05.054. Epub 2016 Jun 18. PMID 27288217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from Italy and Sweden were randomized to Rotavirus Vaccine Subset 1 (Rotarix™). Participants from Finland were randomized to Rotavirus Vaccine Subset 2 (RotaTeq™).
Period: Infant Series
Arm/Group | PR5I | INFANRIX™ Hexa
Started | 656 | 659
Vaccinated | 653 | 659
Completed | 649 | 651
Not Completed | 7 | 8
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Not Vaccinated | 3 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 6
Period: Interim Period
Arm/Group | PR5I | INFANRIX™ Hexa
Started | 649 | 651
Completed | 639 | 642
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 9 | 6
Period: Toddler Dose
Arm/Group | PR5I | INFANRIX™ Hexa
Started | 639 | 642
Completed | 639 | 642
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PR5I | INFANRIX™ Hexa | Total
Number analyzed (Participants) | 656 | 659 | 1315
Age, Continuous [Mean (Standard Deviation); unit: Days] | 68 (10.3) | 68.1 (10.5) | 68.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 323 | 313 | 636
  Male | 333 | 346 | 679
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 459 | 460 | 919
  Italy | 132 | 132 | 264
  Sweden | 65 | 67 | 132

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Antibody (Ab) Response or Seroresponse Rates to All Antigens Contained in PR5I Vaccine One Month After the Toddler Dose of PR5I (11 to 12 Months of Age)
Description: Acceptability response rates were defined as Ab titre ≥1.0 μg/mL for Haemophilus influenzae type b (Hib) (polyribosylribitol phosphate, PRP); ≥10 mIU/mL for Hepatitis (HBsAg); ≥0.1 IU/mL for diphtheria and tetanus; ≥8 (1/dil) for inactive poliovirus type (IPV) 1, 2 & 3, and percentage of pertussis seroresponder participants (Pertussis toxoid [PT], Filamentous haemagglutinin [FHA], Fimbriae types 2 & 3 [FIM] and Pertactin [PRN]) 1 month Post-Toddler dose of PR5I. Seroresponse was defined: (1) If pre-Dose 1 Ab concentration (cc) was <LLOQ (lower limit of quantitation), postvaccination Ab cc was ≥LLOQ, (2) If pre-Dose 1 Ab cc was ≥LLOQ, postvaccination Ab cc was ≥prevaccination levels. Due to the timing of the occurrence of protocol violation or the availability of each antigen serology testing result, the analysis populations may not have been identical for each antigen-specific analysis at each post-vaccination visit.
Time Frame: 1 month after Toddler dose of PR51 (post-toddler dose)
Population: Participants who met the inclusion criteria, were not protocol violators, received PR51 vaccinations within acceptable day ranges, and had a blood draw sample window of Days 28 to 51 following the Toddler dose. Participants receiving INFANRIX™ hexa were excluded from the acceptability analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 638 | 0
Percentage of participants
  Anti-PRP ≥1.0 μg/mL: number analyzed (Participants) | 454 | 0
  Anti-PRP ≥1.0 μg/mL | 89.87 [86.72 to 92.49] |
  Anti-HBsAg ≥10 mIU/mL: number analyzed (Participants) | 377 | 0
  Anti-HBsAg ≥10 mIU/mL | 98.14 [96.21 to 99.25] |
  Anti-Diphtheria ≥0.1 IU/mL: number analyzed (Participants) | 590 | 0
  Anti-Diphtheria ≥0.1 IU/mL | 98.64 [97.35 to 99.41] |
  Anti-Tetanus ≥0.1 IU/mL: number analyzed (Participants) | 589 | 0
  Anti-Tetanus ≥0.1 IU/mL | 99.83 [99.06 to 100.00] |
  Anti-PT seroresponse: number analyzed (Participants) | 566 | 0
  Anti-PT seroresponse | 99.12 [97.95 to 99.71] |
  Anti-FHA seroresponse: number analyzed (Participants) | 582 | 0
  Anti-FHA seroresponse | 97.42 [95.78 to 98.55] |
  Anti-FIM seroresponse: number analyzed (Participants) | 581 | 0
  Anti-FIM seroresponse | 98.28 [96.86 to 99.17] |
  Anti-PRN seroresponse: number analyzed (Participants) | 582 | 0
  Anti-PRN seroresponse | 96.91 [95.16 to 98.16] |
  Anti-IPV1 ≥1:8 dilution: number analyzed (Participants) | 591 | 0
  Anti-IPV1 ≥1:8 dilution | 99.32 [98.28 to 99.82] |
  Anti-IPV2 ≥1:8 dilution: number analyzed (Participants) | 591 | 0
  Anti-IPV2 ≥1:8 dilution | 99.83 [99.06 to 100.00] |
  Anti-IPV3 ≥1:8 dilution: number analyzed (Participants) | 590 | 0
  Anti-IPV3 ≥1:8 dilution | 99.49 [98.52 to 99.90] |
Statistical Analysis 1: Comparison: PR5I; Anti-PRP ≥ 1.0 μg/mL; Test type: Other — The immune response to PR5I vaccine was considered as acceptable if the lower bounds of the 2-sided 95% CI for the response rates were greater than 75%; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 2: Comparison: PR5I; Anti-HBsAg ≥10 mIU/mL; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 3: Comparison: PR5I; Anti-Diphtheria ≥0.1 IU/mL; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 4: Comparison: PR5I; Anti-Tetanus ≥0.1 IU/mL; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 5: Comparison: PR5I; Anti-PT seroresponse; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 6: Comparison: PR5I; Anti-FHA seroresponse; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 7: Comparison: PR5I; Anti-FIM seroresponse; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 8: Comparison: PR5I; Anti-PRN seroresponse; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 9: Comparison: PR5I; Anti-IPV1 ≥1:8 dilution; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 10: Comparison: PR5I; Anti-IPV2 ≥1:8 dilution; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value
Statistical Analysis 11: Comparison: PR5I; Anti-IPV3 ≥1:8 dilution; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Clopper and Pearson — One-sided p-value

2. Secondary Outcome: Non-inferiority of Antibody (Ab) Response Rate to Haemophilus Influenzae Type b (PRP) One Month After the 2nd Dose of PR5I (4 Months of Age) as Compared With INFANRIX Hexa
Description: Percentage of participants with an Ab titre ≥1.0 μg/mL for Hib (polyribosylribitol phosphate, PRP) measured by radioimmunoassay (RIA) 1 month post-infant dose 2 of PR5I or INFANRIX hexa.
Time Frame: 1 month after the 2nd dose (post-infant dose 2)
Population: Participants who received 2nd dose in the Infant series and had a blood draw sample window of Days 28 to 51 post-infant dose 2.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 609 | 592
Percentage of participants | 72.86 | 26.66
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Test type: Non-Inferiority — If the lower bound of the 95% confidence interval (CI) was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen — Stratification by country; Difference in percentages = 46.20, 95% CI 2-sided [41.05 to 51.06]

3. Secondary Outcome: Superiority of Antibody (Ab) Response Rates to Haemophilus Influenzae Type b (PRP) One Month After the 2nd Dose of PR5I (4 Months of Age) as Compared With INFANRIX Hexa
Description: Percentage of participants with an Ab titre ≥1.0 μg/mL for Hib (polyribosylribitol phosphate, PRP) measured by RIA 1 month post-infant dose 2 of PR5I or INFANRIX hexa.
Time Frame: 1 month after the 2nd dose (post-infant dose 2)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 609 | 592
Percentage of participants | 72.86 | 26.66
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Test type: Superiority — If the lower bound of the 95% CI was greater than 0, it was concluded that PR5I group response rate was superior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen; Stratification by country; Difference in percentages = 46.20, 95% CI 2-sided [41.05 to 51.06]

4. Secondary Outcome: Non-inferiority Ab Response Rates to PR5I Antigens One Month After the Toddler Dose of PR5I (11 to 12 Months of Age) as Compared With INFANRIX Hexa
Description: Percentage of participants with pre-specified Ab titre for PRP, HBsAg, diphtheria, tetanus, IPV1, 2 & 3, and percentage of pertussis seroresponder participants (PT, FHA, FIM and PRN) 1 month post-toddler dose were calculated based on the method by Miettinen and Nurminen stratified by country. Seroresponse was defined: (1) If pre-Dose 1 Ab cc was <LLOQ, post-vaccination Ab cc was ≥LLOQ, (2) If pre-Dose 1 Ab cc was ≥LLOQ, post-vaccination Ab cc was ≥pre-vaccination levels. Due to the timing of the occurrence of protocol violation or the availability of each antigen serology testing result, the analysis populations may not have been identical for each antigen-specific analysis at each post-vaccination visit.
Time Frame: 1 month after Toddler dose (post-toddler dose)
Population: Participants who met the inclusion criteria, were not protocol violators, received vaccinations within acceptable day ranges, and had a blood draw sample window of Days 28 to 51 following the Toddler dose.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 638 | 642
Percentage of participants
  Anti-PRP ≥1.0 μg/mL: number analyzed (Participants) | 454 | 478
  Anti-PRP ≥1.0 μg/mL | 89.80 | 91.06
  Anti-HBsAg ≥10 mIU/mL: number analyzed (Participants) | 377 | 391
  Anti-HBsAg ≥10 mIU/mL | 98.14 | 98.73
  Anti-Diphtheria ≥0.1 IU/mL: number analyzed (Participants) | 590 | 578
  Anti-Diphtheria ≥0.1 IU/mL | 98.62 | 99.83
  Anti-Tetanus ≥0.1 IU/mL: number analyzed (Participants) | 589 | 577
  Anti-Tetanus ≥0.1 IU/mL | 99.83 | 100.00
  Anti-PT seroresponse: number analyzed (Participants) | 566 | 561
  Anti-PT seroresponse | 99.11 | 99.64
  Anti-FHA seroresponse: number analyzed (Participants) | 582 | 571
  Anti-FHA seroresponse | 97.40 | 99.13
  Anti-PRN seroresponse: number analyzed (Participants) | 582 | 572
  Anti-PRN seroresponse | 96.86 | 98.28
  Anti-IPV1 ≥1:8 dilution: number analyzed (Participants) | 591 | 580
  Anti-IPV1 ≥1:8 dilution | 99.32 | 99.83
  Anti-IPV2 ≥1:8 dilution: number analyzed (Participants) | 591 | 579
  Anti-IPV2 ≥1:8 dilution | 99.83 | 100.00
  Anti-IPV3 ≥1:8 dilution: number analyzed (Participants) | 590 | 579
  Anti-IPV3 ≥1:8 dilution | 99.49 | 99.65
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Non-inferiority for PRP; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in PRP response rate (based on Ab titre ≥1.0 μg/mL) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -1.27, 95% CI 2-sided [-5.13 to 2.52]
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for HBsAg; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in HBsAg response rate (based on Ab titre ≥10 mIU/mL) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; ifference in percentages = -0.59, 95% CI 2-sided [-2.66 to 1.35]
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for Diptheria; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in Diphtheria response rate (based on Ab titre ≥0.1 IU/mL) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -1.21, 95% CI 2-sided [-2.54 to -0.22]
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for Tetanus; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in Tetanus response rate (based on Ab titre ≥0.1 IU/mL) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -5% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -0.17, 95% CI 2-sided [-0.95 to 0.50]
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for PT; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in the percentage of seroresponder participants for PT was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -0.54, 95% CI 2-sided [-1.75 to 0.49]
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for FHA; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in the percentage of seroresponder participants for FHA was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -1.73, 95% CI 2-sided [-3.47 to -0.26]
Statistical Analysis 7: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for PRN; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in the percentage of seroresponder participants for PRN was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -10% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -1.42, 95% CI 2-sided [-3.42 to 0.39]
Statistical Analysis 8: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for IPV1; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in IPV1 response rate (based on Ab titre ≥8 (1/dil)) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -5% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -0.51, 95% CI 2-sided [-1.59 to 0.34]
Statistical Analysis 9: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for IPV2; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in IPV2 response rate (based on Ab titre ≥8 (1/dil)) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -5% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -0.17, 95% CI 2-sided [-0.96 to 0.49]
Statistical Analysis 10: Comparison: PR5I vs INFANRIX™ Hexa; Non-Inferiority for IPV3; Test type: Non-Inferiority — The estimate of the difference between PR5I & INFANRIX hexa groups in IPV3 response rate (based on Ab titre ≥8 (1/dil)) was calculated with its 1-sided P-value & 2-sided 95% CI. If the lower bound of the 95% CI was greater than -5% (non-inferiority margin), it was concluded that PR5I group response rate was non-inferior to INFANRIX hexa group response rate; p < 0.001, Miettinen & Nurminen with stratification; Statistical analysis was based on the Miettinen & Nurminen method stratified by country; Difference in percentages = -0.16, 95% CI 2-sided [-1.20 to 0.82]

5. Secondary Outcome: Non-inferiority of Rotavirus Response (Geometric Mean Titer, GMT) One Month After the 2nd Dose of Rotarix (4 Months of Age) Administered Concomitantly With PR5I Versus INFANRIX Hexa
Description: Antibody titres expressed in units/mL were measured for Rotavirus IgA by Enzyme Immunoassay (EIA), 1 month after the 2nd dose of Rotarix, administered concomitantly with PR5I or INFANRIX hexa (Post-Dose 2). The 95% CI for GMT was based on the t-distribution of the natural log-transformed antibody titer.
Time Frame: 1 month after the 2nd dose of Rotarix, administered concomitantly with PR5I or INFANRIX hexa (Post-Dose 2)
Population: Participants who received dose 2 of Rotarix.
Measure: Geometric Mean (95% Confidence Interval); unit: Titre (units/mL)
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 160 | 171
Titre (units/mL) | 96.41 [71.69 to 129.65] | 122.24 [92.48 to 161.58]
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Test type: Non-Inferiority — The estimate for anti-rotavirus IgA GMT ratio (PR5I group/INFANRIX hexa group) was calculated with its 1-sided P-value and 2-sided 95% CI. If the lower bound of the 95% CI for GMT ratio was greater than 0.50 (non-inferiority margin), it was concluded that the Rotarix antigen response in the PR5I group was not inferior to the Rotarix antigen response in the INFANRIX hexa group; p = 0.011, ANCOVA; Geometric Mean Titre (GMT) ratio = 0.80, 95% CI 2-sided [0.54 to 1.20]

6. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE) From Day 1 to Day 15 After Any Vaccination
Description: Injection-site and systemic AEs were reported daily on the Vaccination Report Card (VRC) by the parent(s) or legal representative from Day 1 (D1) to D15 after each vaccination. Solicited injection site and systemic AEs were reported daily from D1 to D5 after each vaccination. AEs at injection sites were always considered as vaccine-related (V-related) (Injection-Site Reactions [ISRs]). The investigator had to assess whether systemic AEs were related or not to the vaccine. All AEs (related and unrelated) are displayed here.
Time Frame: Solicited AEs: up to 5 days (Days 1-5 after any vaccination); unsolicited AEs: up to 15 days (Day 1-15 after any vaccination)
Population: All randomized participants who received at least 1 vaccination and who had safety follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 653 | 659
Percentage of participants
  At least 1 ISR or systemic AE (D1-D15) | 99.5 | 99.2
  At least 1 ISR or V-related systemic AE (D1-D15) | 99.5 | 98.8
  At least 1 ISR (D1-D15) | 90.8 | 88.2
  At least 1 solicited ISR (D1-D5) | 90.4 | 87.9
  At least 1 systemic AE (D1-D15) | 99.1 | 98.9
  At least 1 V-related systemic AE (D1-D15) | 99.1 | 98.3
  At least 1 solicited systemic AE (D1-D5) | 99.1 | 98.3
  At least 1 V-related solicited systemic AE (D1-D5) | 99.1 | 98.2
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; ISR or systemic AE; Test type: Other — The risk differences between groups (PR5I group - INFANRIX hexa group) and their 2-sided 95% CI were calculated for the above criteria based on the unstratified Miettinen & Nurminen method. The aim of the 95% CI was to investigate an overall trend and not any specific difference. If 0.0 was excluded from the 95% CI, the trend could not be ruled out; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.7 to 1.4]
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; ISR or V-related systemic AE; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.8, 95% CI [-0.3 to 2.0]
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; At least 1 ISR; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 2.6, 95% CI 2-sided [-0.7 to 6.0]
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; At least 1 solicited ISR; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 2.5, 95% CI 2-sided [-0.9 to 5.9]
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; At least 1 systemic AE; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.1, 95% CI 2-sided [-1.1 to 1.4]
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; At least 1 vaccine-related systemic AE; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-0.5 to 2.2]
Statistical Analysis 7: Comparison: PR5I vs INFANRIX™ Hexa; At least 1 solicited systemic AE; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-0.5 to 2.2]
Statistical Analysis 8: Comparison: PR5I vs INFANRIX™ Hexa; At least 1 vaccine-related solicited systemic AE; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.9, 95% CI [-0.4 to 2.3]

7. Secondary Outcome: Percentage of Participants Reporting Solicited ISRs From D1 to D5 After Any Vaccination
Description: Adverse events at injection sites were always considered as related to vaccine (Injection-Site Reactions [ISRs]). Solicited ISRs were defined as injection-site erythema, injection-site pain, and injection-site swelling occurring from D1 to D5 after vaccination.
Time Frame: Up to 5 days (Day 1 to Day 5 following vaccination)
Population: All randomised participants who received at least 1 vaccination and who had safety follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 653 | 659
Percentage of participants
  Injection-site erythema | 68.6 | 60.4
  Injection-site pain | 73.4 | 70.0
  Injection-site swelling | 56.8 | 49.3
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site erythema; Test type: Other — The risk differences between groups (PR5I group - INFANRIX hexa group) and their 2-sided 95% CI were calculated for the above criteria based on the unstratified Miettinen & Nurminen method. The aim of the 95% CI was to investigate whether an overall trend of risk differences existed. If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; Risk Difference (RD) = 8.2, 95% CI 2-sided [3.0 to 13.3]
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site pain; Test type: Other — [test comment as in outcome 7, analysis 1]; Risk Difference (RD) = 3.4, 95% CI 2-sided [-1.5 to 8.3]
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site swelling; Test type: Other — [test comment as in outcome 7, analysis 1]; Risk Difference (RD) = 7.5, 95% CI [2.1 to 12.9]

8. Secondary Outcome: Percentage of Participants Reporting Unsolicited ISRs From D1 to D15 After Any Vaccination
Description: Adverse events at injection sites were always considered as related to vaccine (Injection-Site Reactions {ISRs]). Unsolicited ISRs occurring from Day 1 (D1) to D15 after any vaccination were reported daily on the VRC by the parent(s) or legal representative. Unsolicited ISRs with incidence ≥1% are reported below.
Time Frame: From D1 to D15 after any vaccination
Population: All randomised participants who received at least 1 vaccination and who had safety follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 653 | 659
Percentage of participants
  Injection-site bruising | 0.9 | 2.0
  Injection-site haemorrhage | 1.8 | 1.8
  Injection-site induration | 15.8 | 13.2
  Injection-site nodule | 1.1 | 0.8
  Injection-site warmth | 2.3 | 1.2
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site bruising; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = -1.1, 95% CI 2-sided [-2.5 to 0.3]
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site haemorrhage; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.5 to 1.6]
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site induration; Test type: Other; Risk Difference (RD) = 2.6, 95% CI 2-sided [-1.2 to 6.4]
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site nodule; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.8 to 1.5]
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Injection-site warmth; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 1.1, 95% CI [-0.4 to 2.7]

9. Secondary Outcome: Percentage of Participants Reporting Solicited Adverse Events (AEs) From D1 to D5 After Any Vaccination
Description: Solicited systemic AEs were defined as crying, decreased appetite, irritability, pyrexia (rectal temperature ≥38.0°C), somnolence, and vomiting occurring from D1 to D5 after vaccination. The investigator had to assess whether these systemic AEs were related or not to the vaccines. All (related and unrelated) are displayed here.
Time Frame: Up to 5 days (from D1 to D5 after any vaccination)
Population: All randomised participants who received at least 1 vaccination and who had safety follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | PR5I | INFANRIX™ Hexa
Number analyzed (Participants) | 653 | 659
Percentage of participants
  Crying | 89.3 | 87.1
  Decreased appetite | 65.8 | 62.2
  Irritability | 91.6 | 89.4
  Pyrexia | 73.8 | 67.4
  Somnolence | 86.1 | 80.3
  Vomiting | 32.8 | 31.0
Statistical Analysis 1: Comparison: PR5I vs INFANRIX™ Hexa; Crying; Test type: Other — [test comment as in outcome 7, analysis 1]; Risk Difference (RD) = 2.2, 95% CI 2-sided [-1.3 to 5.7]
Statistical Analysis 2: Comparison: PR5I vs INFANRIX™ Hexa; Decreased appetite; Test type: Other — The risk differences between groups (PR5I group - INFANRIX hexa group) and their 2-sided 95% CI were calculated for the above criteria based on the unstratified Miettinen & Nurminen method. If the 95% CI for the risk differences included 0.0, the numerical differences were not considered significant; Risk Difference (RD) = 3.6, 95% CI 2-sided [-1.6 to 8.8]
Statistical Analysis 3: Comparison: PR5I vs INFANRIX™ Hexa; Irritability; Test type: Other — [test comment as in outcome 9, analysis 2]; Risk Difference (RD) = 2.2, 95% CI 2-sided [-1.0 to 5.4]
Statistical Analysis 4: Comparison: PR5I vs INFANRIX™ Hexa; Pyrexia; Test type: Other — [test comment as in outcome 9, analysis 2]; Risk Difference (RD) = 6.4, 95% CI 2-sided [1.5 to 11.3]
Statistical Analysis 5: Comparison: PR5I vs INFANRIX™ Hexa; Somnolence; Test type: Other — [test comment as in outcome 6, analysis 1]; Risk Difference (RD) = 5.8, 95% CI 2-sided [1.7 to 9.8]
Statistical Analysis 6: Comparison: PR5I vs INFANRIX™ Hexa; Vomiting; Test type: Other — [test comment as in outcome 9, analysis 2]; Risk Difference (RD) = 1.8, 95% CI 2-sided [-3.2 to 6.9]

ADVERSE EVENTS:
Time Frame: Up to approximately 11 months (serious AEs and deaths were collected for the duration of the study; unsolicited adverse events were collected from D1 to D15 after each hexavalent vaccination, solicited adverse events were collected D1 to D5 after each hexavalent vaccination)
Description: Analysis population includes all randomised participants who received at least 1 vaccination and had safety follow-up.
Arm/Group | PR5I | INFANRIX™ Hexa
All-Cause Mortality (participants affected / at risk) | 0/653 | 0/659
Serious Adverse Events (participants affected / at risk) | 6/653 | 10/659
Other Adverse Events (participants affected / at risk) | 650/653 | 653/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR5I (N=653) | INFANRIX™ Hexa (N=659)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR5I (N=653) | INFANRIX™ Hexa (N=659)
Abdominal pain (Gastrointestinal disorders) | 20 (23) | 10 (11)
Constipation (Gastrointestinal disorders) | 22 (25) | 16 (18)
Diarrhoea (Gastrointestinal disorders) | 76 (95) | 70 (84)
Flatulence (Gastrointestinal disorders) | 29 (32) | 25 (29)
Vomiting (Gastrointestinal disorders) | 220 (324) | 211 (319)
Crying (General disorders) | 583 (1422) | 574 (1305)
Injection site bruising (General disorders) | 13 (15) | 23 (24)
Injection site erythema (General disorders) | 485 (1625) | 450 (1490)
Injection site haemorrhage (General disorders) | 17 (21) | 17 (20)
Injection site induration (General disorders) | 119 (266) | 107 (246)
Injection site pain (General disorders) | 496 (1778) | 493 (1656)
Injection site swelling (General disorders) | 406 (1179) | 373 (1083)
Irritability (General disorders) | 598 (1518) | 589 (1446)
Pyrexia (General disorders) | 490 (875) | 452 (768)
Nasopharyngitis (Infections and infestations) | 35 (39) | 36 (39)
Otitis media (Infections and infestations) | 24 (26) | 15 (15)
Rhinitis (Infections and infestations) | 34 (39) | 41 (44)
Upper respiratory tract infection (Infections and infestations) | 41 (45) | 43 (48)
Decreased appetite (Metabolism and nutrition disorders) | 431 (731) | 411 (694)
Somnolence (Nervous system disorders) | 562 (1168) | 529 (1118)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 24 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor and Sponsor representative must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor or Sponsor representative as confidential must be deleted prior to submission.